CLINICAL TRIAL: NCT05787080
Title: The Effect of Massage on Oxidative and Antioxidant Enzymes in Hemodialysis Patients With Restless Legs Syndrome
Brief Title: Massage, Oxidative and Antioxidant Enzymes in Hemodialysis Patients With Restless Legs Syndrome(RLS)
Acronym: RLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Gülay Turgay, assistant professor, Baskent University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: G Turgay
Record Dates: First submitted 2023-02-06; First posted 2023-03-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-01

CONDITIONS: Renal Failure Chronic; Restless Legs Syndrome
Keywords: renal failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Restless Legs Syndrome; Renal Insufficiency | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Massage/experimental Group- control Group
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcomes assessor will not be in the control and experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Group/experimental (Experimental): Blood tests will be taken at the entrance of dialysis from all participants. Then, in the second hour of hemodialysis, low voltage vibrations will be applied to both calf muscles of the patients for 10 minutes, three times a week for one month.Vibration application will be made with this device 53 Hz head. The vibration application will be performed for 2.5 minutes, starting from the medial side of the gastrocnemius (calf) muscle in both legs and moving it longitudinally from distal to proximal and from back to distal in a straight line within 20 seconds. Then this treatment will be applied to the lateral side of the gastrocnemius muscle for 2.5 minutes. This cycle will be repeated twice. After the one-month application period is completed, blood tests will be taken from all participants at the entrance to hemodialysis.
  Interventions: Other: Massage
- Control Group (No Intervention): No intervention will be made on the patients in the control group.

INTERVENTIONS:
Other: Massage — In the second hour of hemodialysis, vibration is applied to both calf muscles of the patients for 10 minutes three times a week for four weeks at low voltages.
  Arms: Massage Group/experimental

SUMMARY:
This study; It will be done to evaluate the presence of oxidative stress and its effects on lipid peroxidation products and antioxidant parameters after massage application and the possible effects of the appropriate massage protocol applied to the patients on oxidative stress in hemodialysis patients with restless legs syndrome.

DETAILED DESCRIPTION:
In this study, the following research hypotheses will be tested. H0a: Individuals with restless legs syndrome receiving hemodialysis treatment; In the second hour of hemodialysis, massage applied to both calf muscles for 10 minutes three times a week for one month is not affect the oxidative and antioxidant enzymes of the patients.

H1a: Individuals with restless legs syndrome receiving hemodialysis treatment; In the second hour of hemodialysis, massage applied to both calf muscles for 10 minutes three times a week for one month is effective on the oxidative and antioxidant enzymes of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving hemodialysis treatment for at least 6 months, 3 days a week for 4 hours,
2. Patients with RLS according to the diagnostic criteria of the International RLS study group,
3. No psychiatric problems,
4. No neurological deficit,
5. Exercise and physical therapy modalities have not been applied in the last year,
6. In the laboratory examinations, the kinetic indicators of dialysis adequacy are within the desired target range (Kt/V: 1.2-1.3; URR: 60-65%), and there are no pathological findings (fracture, dislocation, tumor, infection) in the radiological examinations. .

Exclusion Criteria:

1. Hemiplegic patients
2. Patients with heart failure
3. Individuals with chronic obstructive pulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) levels of RLS patients | 1 week
  In patients diagnosed with RLS, their blood will be taken on the same day and their plasma will be collected by centrifugation. In RLS patients, cells are expected to undergo lipid peroxidation depending on the disease. This causes cell and tissue damage due to oxidative stress. Damage can also increase the severity and extent of the pain. For this reason, the degree of degradation will be determined by measuring the color reaction-based concentration (nmol/ml plasma) formed as a result of the reaction of malondialdehyde, the degradation product of lipids, which is an indicator of lipid peroxidation, with thiobarbituric acid (TBA).
Erythrocyte Reducte Glutathione (GSH) levels of RLS patients | 1 week
  Reduced glutathione is needed to stay healthy and prevent disease and protect from the effects of aging, immune function and control of inflammation. After adding an equal amount of 10% TCA to plasma samples from 24 RLS patients. It was centrifuged at 4000 rpm at +4ºC for 10 minutes. 0.5 ml of the upper phase is taken and 2 ml of 0.3 M Na2HPO4, 2H2O and 0.2 ml of dithiobisnitro benzoic acid are added on it, and then 412 nm. will be read in the spectrophotometer and their concentrations will be given in terms of micromole (µmol) / ml plasma. This will also confirm the concentration of lipid peroxidation present.

SECONDARY OUTCOMES:
Effect of vibration massage on blood level of Malondialdehyde | 1 week
  It is expected that a decrease in the concentration of MDA and an increase in the rate of reduced glutathione (GSH) are expected, since it is thought that the vibration vibration massage applied to the same patients may cause the intercellular fluid and blood mobilization due to heat and vibration on the muscle tissue, thereby lowering the pain threshold.
Effect of vibration massage on blood level of Erythrocyte Reducte Glutathione | 1 week
  It is expected that a decrease in the concentration of MDA and an increase in the rate of reduced glutathione (GSH) are expected, since it is thought that the vibration vibration massage applied to the same patients may cause the intercellular fluid and blood mobilization due to heat and vibration on the muscle tissue, thereby lowering the pain threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided